CLINICAL TRIAL: NCT05553756
Title: Impact of Maltodextrin, Given 2 Hours Before Cesarean Section, on Glycemic and Hemodynamic Management of Pregnant
Brief Title: Impact of Maltodextrin on Glycemic and Hemodynamic Management During Cesarean Section
Acronym: MALTO-TC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Foggia (Other)
Collaborators: Casa Sollievo della Sofferenza IRCCS (Other)
Responsible Party: Principal Investigator, Cotoia Antonella, Clinical Professor, University of Foggia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 08/CE
Record Dates: First submitted 2022-03-31; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative clear liquid (No Intervention): Patients will drink 200 ml of clear liquid two hours before Cesarean section
- preoperative maltodextrin (Active Comparator): Patients will drink 200 ml of maltodexin two hours before Cesarean section
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Maltodextrin — 200 ml maltodextrin given 2 hours before cesarean section
  Arms: preoperative maltodextrin

SUMMARY:
The goal is to evaluate the glycemic and hemodynamic stability in patients undergoing caesarean section in patients treated with maltodextrins two hours before the cesarean section

DETAILED DESCRIPTION:
The patients undergoing elective cesarean section will be randomly divided in two groups: patients who drink 200 ml of clear liquid two hours before surgery or patients treated with 200 ml maltodextrins two hours before the surgery. The glycemic control will be done immediately before the maldodextrin administration and after the cesarean section by gluco stick. Standard hemodynamic monitoring ECG, Heart Rate, Blood pressure, Temperature, preipheral oxygen saturation will be done routinely.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* first cesarean section
* single fetus
* ASA I-II

Exclusion Criteria:

* BMI<18
* BMI>35
* contraindication to spinal anesthesia
* cardiovascular diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant
Enrollment: 40 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic stability | perioperative
  blood glucose levels <180 mg/dl
hemodynamic stability | perioperative
  mean arterial pressure > 70 mmHg during perioperative time

CONTACTS AND LOCATIONS:
Locations (1):
- University of Foggia, Foggia, Italy